CLINICAL TRIAL: NCT06529120
Title: Adaptation and Pilot Testing of a Mindfulness-Based Insomnia and Symptom Management Intervention for Women With Breast Cancer Receiving Treatment in Rural Medically Underserved Areas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00116035; 5P30CA014236-50 (NIH)
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nite2Day (Experimental): Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills (Nite2Day)
  The Nite2Day intervention will train participants in mindfulness-based sleep strategies and behavioral symptom management techniques. The Nite2Day intervention will consist of 6 weekly sessions that will between 45 and 60 minutes.
  Interventions: Behavioral: Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills

INTERVENTIONS:
Behavioral: Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills — Mindfulness-based sleep strategies and cognitive-behavioral symptom coping skills.

SUMMARY:
Women with breast cancer often experience multiple difficult symptoms, for example insomnia, fatigue, stress, and pain. This study is being done to test a mindfulness-based insomnia and symptom management intervention for women with breast cancer (Nite2Day). Participants will complete six, 45-60 minute intervention sessions with a study therapist. Intervention sessions will be conducted remotely via conference (i.e., Zoom) or telephone. During these sessions, participants will learn mindfulness and cognitive-behavioral strategies to cope with nighttime sleep disturbances and daytime symptoms of fatigue, stress, and pain. Participants will be asked to complete three, brief (15-20 minute) surveys that will ask questions about their background, cancer diagnosis and treatments, cancer symptoms, and experience with the intervention. Participants will be compensated for completing all intervention sessions and surveys. Total study duration is about 12 weeks.

The greatest risk of this study is loss of confidentiality. Benefits from participating might include learning skills to reduce nighttime sleep disturbances and daytime symptoms of fatigue, stress, and pain. Information learned from this study may also benefit other patients with cancer in the future.

ELIGIBILITY:
Inclusion Criteria:

1. stage 0-IV breast cancer diagnosis within past 12 months
2. self-report >8 on the Insomnia Severity Index, indicating at least mild symptoms of clinical insomnia
3. >18 years old
4. life expectancy of >12 months per medical chart or oncologist
5. Ability to speak and read English, and intact hearing and vision

Exclusion Criteria:

1. reported or suspected cognitive impairment confirmed via Folstein Mini-Mental Status Exam <25;
2. serious psychiatric (e.g., schizophrenia, suicidal intent) or medical condition (e.g., seizure disorder, narcolepsy, severe or moderate untreated sleep apnea) indicated by self-report, medical chart, or oncologist/provider that would contraindicate safe participation;
3. engagement in behavioral insomnia (e.g., Cognitive-Behavioral Therapy for Insomnia) or symptom management (e.g., Pain Coping Skills Training) interventions within past 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility as measured by study accrual | 6 months of study recruitment
  Treatment feasibility will be shown by meeting targeted study accrual (N = 15) in 6 months
Feasibility as measured by study attrition | 12 weeks (post-intervention)
  Treatment feasibility will be shown by no more than 25% study attrition
Feasibility as measured by adherence | 16 weeks (1-month post-intervention)
  Adherence will be indicated by at least 75% of participants completing all study sessions and assessments
Acceptability as measured by the 10-item Client Satisfaction Questionnaire (CSQ) | 12 weeks (post-intervention)
  Acceptability will be indicated by at least 80% of the participants reporting satisfaction with the protocol on the CSQ. Items are rated on a 4-point scale from 1 (low) to 4 (high) and averaged to obtain an acceptability score ranging from 1 to 4, with higher scores indicating higher acceptability.
Change in insomnia symptoms | 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
  Insomnia symptoms will be measured using the 7-item Insomnia Symptom Index (ISI). Items are summed to yield a total score ranging from 0 to 28, with higher scores indicating worse insomnia symptoms.

SECONDARY OUTCOMES:
Change in fatigue symptoms | 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
  Fatigue symptoms will be assessed using the 8-item PROMIS Fatigue Short Form. A raw score is calculated by summing all 8 items, yielding a total raw score that ranges from 8 to 40. The total raw score is then translated to a T-score, which is a standardized score with a mean of 50 and a standard deviation of 10. Higher T-scores indicated higher fatigue.
Change in depressive symptoms | 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
  Depressive symptoms will be assessed using the 8-item PROMIS Depression Short Form. A raw score is calculated by summing all 8 items, yielding a total raw score that ranges from 8 to 40. The total raw score is then translated to a T-score, which is a standardized score with a mean of 50 and a standard deviation of 10. Higher T-scores indicate higher worse depressive symptoms.
Change in anxiety symptoms | 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
  Anxiety symptoms will be assessed using the 8-item PROMIS Anxiety Short Form. A raw score is calculated by summing all 8 items, yielding a total raw score that ranges from 8 to 40. The total raw score is then translated to a T-score, which is a standardized score with a mean of 50 and a standard deviation of 10. Higher T-scores indicate worse anxiety symptoms.
Change in pain severity | 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
  Pain severity will be assessed using the 11-item Brief Pain Inventory-Short Form (BPI-SF). The BPI-SF consists of 4 items assessing pain severity, including worst, least, average, and current pain in the past week. Responses range from 0 (no pain) to 10 (pain as bad as you can imagine); items are averaged for a composite score that ranges from 0 to 10 with higher scores indicating high pain severity.
Change in pain interference | 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
  Pain interference will be assessed using the 11-item Brief Pain Inventory-Short Form (BPI-SF). The BPI-SF consists of 7 items assessing the degree to which pain has interfered with patients' daily activities in the past week. Responses range from 0 (does not interfere) to 10 (completely interferes); items are averaged for a composite score that ranges from 0 to 10 with higher scores indicating high pain interference.
Change in mindfulness | 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
  Mindfulness will be assessed using the 10-item Cognitive and Affective Mindfulness Scale - Revised (CAMS-R). Items are summed to achieve a total score ranging from 10 to 40. Higher scores indicate higher levels of mindfulness.
Change in self-efficacy for symptom management | 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
  Self-efficacy for symptom management will be measured using the 8-item PROMIS Self-Efficacy for Managing Chronic Conditions (Managing Symptoms) measure. A raw score is calculated by summing all 8 items, yielding a total raw score that ranges from 8 to 40. The total raw score is then translated to a T-score, which is a standardized score with a mean of 50 and a standard deviation of 10. Higher T-scores indicate higher self-efficacy for managing chronic conditions (managing symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Hannah M Fisher, PhD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Calvert Health System, Prince Frederick, Maryland
  - Duke Lifepoint Hospital Maria Parham Medical Center, Henderson, North Carolina
  - Scotland Health Care System, Laurinburg, North Carolina
  - UNC Health Johnston, Smithfield, North Carolina

IPD SHARING:
Plan to Share IPD: No